CLINICAL TRIAL: NCT02101151
Title: Effect of Vitamin D Supplementation on the Metabolic Control and Body Composition of Type 2 Diabetes Subjects in Ajman (UAE)
Acronym: VDIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rashid Centre for Diabetes and Research (Other)
Responsible Party: Principal Investigator, Dr.Amena Sadiya, Senior Nutritionist, Rashid Centre for Diabetes and Research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VDIS
Record Dates: First submitted 2014-03-26; First posted 2014-04-02 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Type 2 Diabetes Mellitus; Obesity; Hypovitaminosis D
Keywords: Type 2 diabetes mellitus; vitamin D; cholecalciferol; obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3 group (Experimental): supplemented with 6000IU cholecalciferol/day for 3 months, followed by 3000 IU cholecalciferol/day for next 3 months
  Interventions: Dietary Supplement: Vitamin D3(cholecalciferol)
- Placebo group (Placebo Comparator): Placebo (starch) capsules identical to vitamin D capsules in appearance
  Interventions: Dietary Supplement: Vitamin D3(cholecalciferol)

INTERVENTIONS:
Dietary Supplement: Vitamin D3(cholecalciferol)
  Other Names: cholecalciferol

SUMMARY:
The incidence of type 2 diabetes mellitus and obesity is increasing at an alarming rate both nationally and worldwide. Accumulating evidence suggests that serum cholecalciferol levels may be inversely related to the prevalence of diabetes, insulin resistance and metabolic syndrome. However, to demonstrate a causal relation between vitamin D and glucose metabolism, evidence from randomized and adequately powered placebo-controlled intervention trials is needed.The trials available on the effect of Vitamin D supplementation are not conclusive. Hence, the purpose of this study was to conduct a double-blind randomized trial in Vitamin D deficient obese type 2 diabetic Emirati population to clarify the effect of vitamin D supplementation on glycemic control and obesity parameters.

DETAILED DESCRIPTION:
Vitamin D insufficiency has been reported as a risk factor for the development of type 1 and type 2 diabetes mellitus. In contrast to the findings of the observational studies, the supplementation trials in type 2 diabetes mellitus (T2DM) do not report any definitive conclusions, but it does suggest that supplementation at an early stage in the development of diabetes may be of benefit in delaying progression to clinical T2DM by increasing the pancreatic insulin release and improved insulin resistance plus impaired glucose tolerance.There is also speculation on role of vitamin D in physiology of weight loss and body composition.However, there have been multiple inconsistencies within the reported trial i.e. sample size, dose of vitamin D, frequency of supplementation, and population studied.

Hence the randomised clinical trial was undertaken to study the effect of vitamin D (Cholecalciferol) supplementation on metabolic markers and obesity parameters in the vitamin D deficient obese type 2 diabetic subjects.

ELIGIBILITY:
Inclusion Criteria:

* United Arab Emirates national
* Male or Female
* Age 30-65 years
* Diagnosed as type 2 diabetes
* Body Mass Index ≥30 kg/m2
* Serum 25 hydroxy Vitamin D ≤ 50nmol/L

Exclusion Criteria:

* Type 1 diabetes mellitus
* History or evidence of liver failure (elevated liver function tests) or renal failure ( elevated creatinine)
* History of malabsorption syndrome.
* On vitamin D Supplementation
* On hormone replacement therapy
* On corticosteroids, anticonvulsants, AIDS medication

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
glycemic control | 6 months
  HbA1c, Fasting Blood glucose, C-peptide

SECONDARY OUTCOMES:
Lipid Profile | 6 months
  Serum Total cholesterol, LDL-C, HDL-C, Triglyceride, Apolipoprotein A and B
Vitamin D | 6 months
  Serum 25-hydroxyvitamin D, Parathyroid hormone, Calcium, Phosphate, Alkaline phosphatase
Other metabolic markers | 6 months
  High sensitive C-Reactive Protein, Creatinine, Thyroid stimulating hormone, Systolic Blood pressure, Diastolic Blood pressure
Obesity Parameter | 6 monhts
  Weight, BMI, waist circumference, Fat mass, Muscle mass, water mass

CONTACTS AND LOCATIONS:
Locations (1):
- Rashid Centre for Diabetes and Research, Ajman, United Arab Emirates

REFERENCES:
- [Derived] Sadiya A, Ahmed SM, Carlsson M, Tesfa Y, George M, Ali SH, Siddieg HH, Abusnana S. Vitamin D3 supplementation and body composition in persons with obesity and type 2 diabetes in the UAE: A randomized controlled double-blinded clinical trial. Clin Nutr. 2016 Feb;35(1):77-82. doi: 10.1016/j.clnu.2015.02.017. Epub 2015 Mar 24. PMID 25892603
- [Derived] Sadiya A, Ahmed SM, Carlsson M, Tesfa Y, George M, Ali SH, Siddieg HH, Abusnana S. Vitamin D supplementation in obese type 2 diabetes subjects in Ajman, UAE: a randomized controlled double-blinded clinical trial. Eur J Clin Nutr. 2015 Jun;69(6):707-11. doi: 10.1038/ejcn.2014.251. Epub 2014 Nov 19. PMID 25406966